CLINICAL TRIAL: NCT00946023
Title: Nonmyeloablative BMT With Post-transplant Cyclophosphamide, Rituximab and Optimized Donor Selection for B-cell Lymphomas
Brief Title: Optimized Donor Selection, Nonmyeloablative BMT for B-cell Lymphomas With Post-transplantation Cy and Rituximab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was unavailable to complete the study as originally planned.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0941; NA_00025589 (Other: Johns Hopkins Medicine Institutional Review Board)
Record Dates: First submitted 2009-07-21; First posted 2009-07-24 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma; B-cell Lymphoma; Non Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: lymphoma; non hodgkin lymphoma; allogeneic; bone marrow transplantation; nonmyeloablative; cyclophosphamide; rituximab
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant (Experimental): Non-myeloablative allogeneic bone marrow transplant (BMT) with a fludarabine (Flu), cyclophosphamide (Cy), total body irradiation (TBI) preparative regimen and post-transplant Cy, mycophenolate mofetil (MMF), and tacrolimus as GVHD (graft vs host disease) prophylaxis. Rituximab will be given as post-transplant maintenance.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total body irradiation; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Rituximab; Biological: Allogeneic Bone Marrow Transplant (BMT)

INTERVENTIONS:
Drug: Fludarabine — Days -6 through -2: 30 mg/m^2 IV daily
  Other Names: Fludara
Drug: Cyclophosphamide — Days -6 and -5: 14.5 mg/kg IV daily; Days 3 and 4: 50 mg/kg IV daily
  Other Names: Cytoxan; CTX; Cy
Radiation: Total body irradiation — Day -1: 200 centigray (cGy) in a single fraction
  Other Names: TBI
Drug: Tacrolimus — Start on Day 5 through Day 180
  Other Names: FK-506; FK506; Prograf
Drug: Mycophenolate Mofetil — Days 5 through 35: 15 mg/kg PO three times daily (max 3 g/day)
  Other Names: MMF; CellCept
Drug: Rituximab — Day 30 and every week after for 8 total doses: 375 mg/m^2 IV
  Other Names: Rituxan
Biological: Allogeneic Bone Marrow Transplant (BMT) — Day 0: Donor bone marrow infusion

SUMMARY:
This phase II trial is studying how well giving fludarabine and cyclophosphamide together with total-body irradiation and rituximab works in treating patients with B-cell lymphoma or chronic lymphocytic leukemia who are undergoing an allogeneic (donor) bone marrow transplant. The type of bone marrow transplant is a less intensive or "mini" transplant using a relative as the bone marrow donor. The donated bone marrow stem cells may replace the patient's immune system cells and help destroy any remaining cancer (graft-versus-tumor effect). Patients undergoing this type of transplant often have more than one relative who could be a donor. The trial is also studying a new way of choosing amongst possible donors which might improve how the rituximab works.

DETAILED DESCRIPTION:
This phase II for relapsed or refractory B-cell malignancies builds on the platform of nonmyeloablative, related-donor, HLA (human leukocyte antigen)-matched or HLA-haploidentical BMT with post-transplantation high-dose cyclosphosphamide administered for prophylaxis of graft-versus-host disease and graft rejection. Rituximab is added to the transplant regimen with the goal of augmenting anti-tumor activity. In patients with B-cell lymphomas, specific polymorphisms in the immunoglobulin Fc receptor have been associated with greater sensitivity to rituximab or rituximab-based therapies, translating in some series into higher response rates and improved progression-free survival. This raises the possibility of selecting donors who carry this permissive polymorphism. This trial identifies and selects donors who have the favorable polymorphism at FcgammaR3A-158, thereby potentially conferring greater sensitivity to rituximab in the host after BMT.

ELIGIBILITY:
Inclusion Criteria:

* Poor-risk CD20+, B-cell lymphoma, as follows:

  * Low grade B-cell lymphoma that has failed at least two prior therapies (excluding single agent rituximab), or undergone histologic conversion (if histologic conversion, PR or CR is required):

    1. Follicular grade 1 or 2 lymphoma
    2. Follicular lymphoma not otherwise specified
    3. Marginal zone (or MALT) lymphoma
    4. Lymphoplasmacytic lymphoma / Waldenstrom's macroglobulinemia
    5. Hairy cell leukemia
    6. Small lymphocytic lymphoma / chronic lymphocytic leukemia (SLL/CLL)
    7. Low grade B-cell lymphoma, unspecified
    8. Nodular lymphocyte-predominant Hodgkin lymphoma
* Poor-risk small lymphocytic lymphoma or chronic lymphocytic leukemia, defined by a 17p deletion, 11q deletion, or histologic conversion (if histologic conversion, PR or CR is required)
* Aggressive B-cell non-Hodgkin's lymphoma that has failed at least one prior regimen of multiagent chemotherapy, is in PR (partial remission) or CR (complete remission), and patient is either ineligible for autologous hematopoietic BMT or autologous BMT is not recommended:

  1. Follicular grade 3 lymphoma
  2. Histoconversion of low-grade B-cell lymphoma (including SLL/CLL) to aggressive B-cell non-Hodgkin's lymphoma
  3. Mantle cell lymphoma
  4. Diffuse large B-cell lymphoma (excluding primary CNS [central nervous system] lymphoma)
  5. "Gray zone" or composite lymphomas with combined features of primary mediastinal large B-cell and Hodgkin's lymphoma
  6. Burkitt's lymphoma/leukemia
  7. Atypical Burkitt's lymphoma/leukemia (high grade B-cell lymphoma, unclassified, including that with features intermediate between Burkitt's and diffuse large B-cell lymphoma)
* Must have a related donor who is at least HLA haploidentical
* Any previous BMT must have occurred at least 3 months prior
* Left ventricular ejection fraction at least 35%
* Bilirubin no more than 3.0 mg/dL (unless due to Gilbert's syndrome), and ALT (alanine aminotransferase) and AST (aspartate aminotransferase) no more than 5 x upper limit of normal
* FEV1 (forced expiratory volume in one second) and FVC (forced vital capacity) at least 40% of predicted
* Absence of uncontrolled infection

Exclusion Criteria:

* More than 20% involvement of bone marrow by chronic lymphocytic leukemia
* Active central nervous system lymphoma
* ECOG (Eastern Cooperative Oncology Group) performance status greater than 1 (2,3, and 4)
* HIV positive
* Pregnant or breastfeeding

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette L Kasamon, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Kanakry JA, Gocke CD, Bolanos-Meade J, Gladstone DE, Swinnen LJ, Blackford AL, Fuchs EJ, Huff CA, Borrello I, Matsui WH, Brodsky RA, Rosner GL, Shanbhag S, Luznik L, Jones RJ, Ambinder RF, Kasamon YL. Phase II Study of Nonmyeloablative Allogeneic Bone Marrow Transplantation for B Cell Lymphoma with Post-Transplantation Rituximab and Donor Selection Based First on Non-HLA Factors. Biol Blood Marrow Transplant. 2015 Dec;21(12):2115-2122. doi: 10.1016/j.bbmt.2015.07.012. Epub 2015 Jul 14. PMID 26183076

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 participants were screen failures and did not proceed on the study.
Groups:
- Transplant: Non-myeloablative bone marrow transplant with a fludarabine (Flu), cyclophosphamide (Cy), total body irradiation (TBI) preparative regimen and post-transplant Cy, mycophenolate mofetil (MMF), and tacrolimus as GVHD prophylaxis. Rituximab will be given as post-transplant maintenance.
  Fludarabine: Days -6 through -2: 30 mg/m^2 IV daily
  Cyclophosphamide: Days -6 and -5: 14.5 mg/kg IV daily; Days 3 and 4: 50 mg/kg IV daily
  Total body irradiation: Day -1: 200 centigray (cGy) in a single fraction
  Tacrolimus: Start on Day 5 through Day 180
  Mycophenolate Mofetil: Days 5 through 35: 15 mg/kg PO three times daily (max 3 g/day)
  Rituximab: Day 30 and every week after for 8 total doses: 375 mg/m^2 IV
Period: Overall Study
Arm/Group | Transplant
Started | 83
Completed | 83
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transplant
Number analyzed (Participants) | 83
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 75]
Age, Customized [Count of Participants; unit: Participants]
  >= 60 years old | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 56
Region of Enrollment [Number; unit: participants]
  United States | 83

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Percentage of participants alive and without relapse or disease progression.
Time Frame: 1 year post-intervention
Population: Populations were analyzed as follows:
  1. All participants
  2. Recipients of haploidentical donors (69 participants)
  3. Recipients of VV, VF, and FF donors (17, 43, and 23 participants, respectively, totaling 83 participants)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants
  All participants | 71 [62 to 82]
  Haploidentical recipients: number analyzed (Participants) | 69
  Haploidentical recipients | 70 [61 to 81]
  VV donor: number analyzed (Participants) | 17
  VV donor | 82 [66 to 100]
  VF donor: number analyzed (Participants) | 43
  VF donor | 70 [56 to 85]
  FF donor: number analyzed (Participants) | 23
  FF donor | 65 [44 to 88]

2. Secondary Outcome: Progression-free Survival
Description: Percentage of participants alive with and without relapse.
Time Frame: 2 years post-intervention
Population: Populations were analyzed as follows:
  All participants Recipients of haploidentical donors (69 participants) Recipients of VV, VF, and FF donors (17, 43, and 23 participants, respectively, totaling 83 participants)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants
  All participants | 60 [52 to 70]
  Haploidentical recipients: number analyzed (Participants) | 69
  Haploidentical recipients | 63 [52 to 76]
  VV donor: number analyzed (Participants) | 17
  VV donor | 68 [48 to 96]
  VF donor: number analyzed (Participants) | 43
  VF donor | 59 [46 to 76]
  FF donor: number analyzed (Participants) | 23
  FF donor | 56 [39 to 81]

3. Secondary Outcome: Overall Survival
Description: Percentage of participants alive.
Time Frame: 1 year post intervention
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants
  All participants | 86 [78 to 93]
  Haploidentical recipients: number analyzed (Participants) | 69
  Haploidentical recipients | 83 [74 to 92]
  VV donor: number analyzed (Participants) | 17
  VV donor | 94 [84 to 100]
  VF donor: number analyzed (Participants) | 43
  VF donor | 86 [76 to 97]
  FF donor: number analyzed (Participants) | 23
  FF donor | 78 [63 to 97]

4. Secondary Outcome: Overall Survival
Description: Percentage of participants alive.
Time Frame: 2 years post intervention
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants
  All participants | 76 [67 to 86]
  Haploidentical recipients: number analyzed (Participants) | 69
  Haploidentical recipients | 73 [63 to 84]
  VV donor: number analyzed (Participants) | 17
  VV donor | 87 [71 to 100]
  VF donor: number analyzed (Participants) | 43
  VF donor | 76 [64 to 90]
  FF donor: number analyzed (Participants) | 23
  FF donor | 69 [52 to 91]

5. Secondary Outcome: Relapse
Description: Percentage of participants alive with relapse or disease progression.
Time Frame: 1 year post intervention
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants
  All participants | 20 [13 to 28]
  Haploidentical recipients: number analyzed (Participants) | 69
  Haploidentical recipients | 20 [11 to 30]
  VV donor: number analyzed (Participants) | 17
  VV donor | 18 [0 to 36]
  VF donor: number analyzed (Participants) | 43
  VF donor | 23 [10 to 36]
  FF donor: number analyzed (Participants) | 23
  FF donor | 17 [1 to 33]

6. Secondary Outcome: Relapse
Description: Percentage of participants alive with relapse or disease progression.
Time Frame: 2 years post intervention
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants
  All participants | 27 [17 to 37]
  Haploidentical recipients: number analyzed (Participants) | 69
  Haploidentical recipients | 23 [13 to 34]
  VV donor: number analyzed (Participants) | 17
  VV donor | 25 [3 to 46]
  VF donor: number analyzed (Participants) | 43
  VF donor | 31 [17 to 45]
  FF donor: number analyzed (Participants) | 23
  FF donor | 22 [4 to 39]

7. Secondary Outcome: Non-relapse Mortality
Description: Percentage of participants who died due to BMT-related reasons.
Time Frame: 1 year post intervention
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants | 8 [2 to 14]

8. Secondary Outcome: Incidence of Grades II-IV Acute Graft-versus-Host-Disease (GVHD)
Description: Percentage of participants who experienced grade II, III, or IV acute GVHD. Acute GVHD is graded using the Przepiorka criteria.
Time Frame: 1 year post intervention
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants | 41 [30 to 52]

9. Secondary Outcome: Incidence of Grades III-IV Acute GVHD
Description: as for outcome 8
Time Frame: 1 year post intervention
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants | 5 [0 to 9]

10. Secondary Outcome: Incidence of Chronic GVHD
Description: Percentage of participants who experienced chronic GVHD. Chronic GVHD is graded using NIH consensus criteria and Seattle criteria.
Time Frame: 1 year post intervention
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants | 11 [4 to 18]

11. Secondary Outcome: Engraftment
Description: Percentage of patients who engrafted neutrophils and platelets.
Time Frame: Day 60
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transplant
Number analyzed (Participants) | 83
percentage of participants
  Neutrophil engraftment | 98 [94 to 100]
  Platelet engraftment | 98 [94 to 100]

12. Secondary Outcome: Graft Failure
Description: Percentage of participants who failed to engraft.
Time Frame: Day 60
Population: Two participants were not analyzed because they died prior to Day 60.
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant
Number analyzed (Participants) | 81
Participants | 2

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were assessed by the investigator and by labwork at each study visit as per protocol.
Arm/Group | Transplant
All-Cause Mortality (participants affected / at risk) | 34/83
Serious Adverse Events (participants affected / at risk) | 56/83
Other Adverse Events (participants affected / at risk) | 62/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant (N=83)
Allergic reaction (Immune system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (2)
Hypotension (Cardiac disorders) | 5 (5)
Tachycardia (Cardiac disorders) | 1 (1)
Rigors/chills (General disorders) | 5 (5)
Dehydration (Gastrointestinal disorders) | 2 (2)
Failure to thrive (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Volume overload (Cardiac disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Cholelithiasis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (9)
Bleeding (Blood and lymphatic system disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 48 (132)
Hyperkalemia (Investigations) | 1 (1)
Hypogammaglobulinemia (Investigations) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Altered consciousness (Nervous system disorders) | 7 (9)
Optic neuritis (Nervous system disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory acidosis (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 8 (8)
Hemophagocytic syndrome (Immune system disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Blood and lymphatic system disorders) | 4 (4)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant (N=83)
Fever (General disorders) | 5 (5)
Infection (Infections and infestations) | 46 (86)
Neutropenic fever (Infections and infestations) | 11 (13)
Neutropenia (Blood and lymphatic system disorders) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 33 (43)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes